CLINICAL TRIAL: NCT05341921
Title: The Acute Effects of Pranayama (Deep Breathing Techniques) on Physiological Parameters in Pregnancy
Brief Title: Deep Breathing Techniques (Pranayama) in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00002180
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy Related; Hypertension in Pregnancy; Blood Pressure
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Intervention Model Description: Pilot, randomized, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Alternate Nostril Breathing Phase I (Active Comparator): Alternate nostril breathing for normotensive women in 3rd trimester of pregnancy
  Interventions: Behavioral: Alternate Nostril Breathing
- Bhramari Breathing Phase I (Active Comparator): Bhramari breathing for normotensive women in 3rd trimester of pregnancy
  Interventions: Behavioral: Bhramari Breathing
- Sheetali Breathing Phase I (Active Comparator): Sheetali breathing for normotensive women in 3rd trimester of pregnancy
  Interventions: Behavioral: Sheetali Breathing
- Alternate Nostril Breathing Phase II (Active Comparator): Alternate nostril breathing for hypertensive women in 3rd trimester of pregnancy
  Interventions: Behavioral: Alternate Nostril Breathing
- Bhramari Breathing Phase II (Active Comparator): Bhramari breathing for hypertensive women in 3rd trimester of pregnancy
  Interventions: Behavioral: Bhramari Breathing
- Sheetali Breathing Phase II (Active Comparator): Sheetali breathing for hypertensive women in 3rd trimester of pregnancy
  Interventions: Behavioral: Sheetali Breathing

INTERVENTIONS:
Behavioral: Alternate Nostril Breathing — Utilizing Pranayama (deep breathing technique) in normotensive and hypertensive women in 3rd trimester of pregnancy
  Arms: Alternate Nostril Breathing Phase I; Alternate Nostril Breathing Phase II
Behavioral: Bhramari Breathing — Utilizing Pranayama (deep breathing technique) in normotensive and hypertensive women in 3rd trimester of pregnancy
  Arms: Bhramari Breathing Phase I; Bhramari Breathing Phase II
Behavioral: Sheetali Breathing — Utilizing Pranayama (deep breathing technique) in normotensive and hypertensive women in 3rd trimester of pregnancy
  Arms: Sheetali Breathing Phase I; Sheetali Breathing Phase II

SUMMARY:
Slow deep breathing actives the vagal nerve and leads to a natural reduction in physiological parameters such as blood pressure, heart rate and digestion. The effects of these techniques have not been assessed in pregnancy. The primary objective is to assess the effects of various yogic deep breathing techniques on blood pressure during pregnancy. The breathing exercises will include Alternate nostril breathing, Bhramari breathing, and Sheetali breathing. A secondary objective will be to assess the effects of these breathing exercises on other physiological parameters including heart rate, heart rate variability, body temperature, cardiac output, vascular resistance and respiratory rate.

DETAILED DESCRIPTION:
The trial will be conducted as a pilot study in one study visit, which will be conducted in two phases. Phase I will be conducted on normotensive pregnant women and Phase II will be conducted on hypertensive pregnant women. Participants will be in their third trimester of pregnancy (28 weeks onwards).

Upon presentation, they will be randomized into one of three groups: Alternate nostril breathing, Bhramari breathing or Sheetali breathing. Maternal monitoring devices will be placed on the patient before the intervention. The fetus will be monitored by external monitors consisting of a fetal heart rate monitor and tocodynamometer to assess uterine activity. Fetal position will be assessed before and after the intervention by ultrasound. All devices will obtain a reading for 15 minutes before, during and after the intervention.

Intervention: In an upright, seated position, the participant will engage in a total of 15 minutes of one deep breathing technique. The breathing practice will be conducted in three, 5-minute increments with a one-minute break between each session. These breathing techniques are easy to learn and participants will be taught how to perform the exercise (visual demonstration, verbal and written instructions will be provided). Participants will be given the opportunity to practice the breathing technique and ask any questions prior to initiating monitoring.

ELIGIBILITY:
Inclusion Criteria:

- Any pregnant woman in the 3rd trimester after 28 weeks of pregnancy who is/has

* 18 years of age or older
* English speaking
* Phase II Only- Chronic hypertension - defined as pre-existing elevated blood pressure prior to pregnancy or less than 20 weeks gestation (Systolic blood pressure greater than or equal to 140 mmHg and /or a diastolic blood pressure greater than or equal to 90 mmHg) with or without antihypertensive use
* Phase II Only- Gestational hypertension - defined as elevated blood pressure (Systolic blood pressure greater than or equal to 140 mmHg and /or a diastolic blood pressure greater than or equal to 90 mmHg) after 20 weeks of pregnancy without any evidence of end-organ damage or proteinuria, with or without antihypertensive use
* Phase II Only- Preeclampsia without severe features - defined as elevated blood pressure (Systolic blood pressure greater than or equal to 140 mmHg but less than 160 mmHG and /or a diastolic blood pressure greater than or equal to 90 mmHg but less than 110 mmHg on two or more occasions 4 hours or more apart) with evidence of proteinuria, with or without antihypertensive use

Exclusion Criteria:

* Any unstable maternal or fetal condition that requires urgent delivery
* Any concerns for pre-eclampsia with or without severe features (i.e. Development of HELLP syndrome or eclampsia)
* Severe pulmonary disease
* Active or acute pulmonary disease
* Known deviated nasal septum
* Does not desire to perform breath-controlled exercises
* Low blood pressure defined as baseline blood pressure less or equal to a systolic of 90 mmHg and/or a diastolic blood pressure of 60 mmHg
* Cannot roll their tongue
* Have difficulty or cannot breathe through their nose

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change of blood pressure from baseline in normotensive and hypertensive women in 3rd trimester pregnancy while utilizing various pranayama breathing techniques | One visit, 15 minute intervention
  Continuous blood pressure monitored while participants engage in a deep breathing technique (pranayama breathing)

SECONDARY OUTCOMES:
Change of heart rate from baseline to after the intervention | One visit, 15 minute intervention
  Continuous heart rate monitor will be applied
Change in body temperature from baseline to after the intervention | One visit, 15 minute intervention
  Continuous temperature monitor will be applied
Change in cardiac output from baseline to after the intervention | One visit, 15 minute intervention
  Continuous cardiac output monitor will be applied

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Babbar, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Advent Health Shawnee Mission Birth Center, Merriam, Kansas, United States

IPD SHARING:
Plan to Share IPD: No